CLINICAL TRIAL: NCT04788745
Title: Targeting Metabolic Flexibility in ALS (MetFlex); Safety and Tolerability of Trimetazidine for the Treatment of ALS
Brief Title: Targeting Metabolic Flexibility in Amyotrophic Lateral Sclerosis (ALS)
Acronym: MetFlex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: FightMND (Other); UMC Utrecht (Other); King's College London (Other); Julius Clinical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MetFlex
Record Dates: First submitted 2021-03-02; First posted 2021-03-09 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2022-11

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Trimetazidine

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm study without placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Trimetazidine 35mg
  Interventions: Drug: Trimetazidine Dihydrochloride

INTERVENTIONS:
Drug: Trimetazidine Dihydrochloride — Oral tablet, twice-daily

SUMMARY:
MetFlex is an investigator led, open-label, single-arm, Phase 2a trial to determine the safety and tolerability of trimetazidine for the treatment of amyotrophic lateral sclerosis/motor neuron disease (ALS/MND).

DETAILED DESCRIPTION:
The study will consist of a 4-week lead-in period to obtain a stable baseline measurement of clinical markers of disease and oxidative stress. After the lead-in phase, participants will receive trimetazidine for 12 weeks. Participants will visit the clinic at 6-week intervals, during which we will obtain a blood sample to measure the pharmacodynamic response. We will also collect information regarding the rate of disease progression (i.e. ALSFRS-R and SVC). At weeks 3 and 9 of treatment, participants will conduct a teleconference visit, during which we will collect data on ALSFRS-R. Adverse events will be collected and recorded throughout the entire trial duration. At the end of the on-treatment period, a close-out visit will occur after four weeks. The total study period per participant will be 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Signed informed consent prior to the initiation of any study-specific procedures
* Familial or sporadic ALS/MND, defined as clinically possible, probable, or definite as per the El Escorial criteria
* Relative TRICALS risk score between -6.0 to -2.0 (75% of patients with ALS/MND)
* Metabolic index ≥110%, at the screening visit.
* The use of riluzole will be permitted during the study. Individuals taking riluzole must be on a stable dose for at least 30 days prior to the baseline visit, or stopped taking riluzole at least 30 days prior to the baseline visit.
* Ability to swallow tablets
* Able to lie with torso elevated at a 35° angle for 30 minutes without respiratory support
* Able to give informed consent (as judged by the investigator) and able to comply with all study visits and all study procedures
* Females must not be able to become pregnant (e.g. post-menopausal, surgically sterile or using highly effective birth control methods) for the duration of the study. Highly effective methods of birth control are those with a failure rate of < 1% per year when employed consistently and correctly, e.g. Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

  * oral
  * intravaginal
  * transdermal
  * Progestogen-only hormonal contraception associated with inhibition of ovulation:
  * oral
  * injectable
  * implantable
  * intrauterine device (IUD)
  * intrauterine hormone-releasing system ( IUS)
  * vasectomised partner
* Females of child-bearing potential must have a negative serum pregnancy test at screening and baseline and be non-lactating

Exclusion Criteria:

* Unable to provide informed consent
* History of, or current diagnosis of diabetes or medical condition that impacts whole body energy expenditure (e.g. Hashimoto's, heart disease)
* Parkinson's disease or parkinsonism, tremor, restless-leg syndrome
* Safety Laboratory Criteria at screening related to significant kidney disease:

  * Creatinine clearance < 50 mL / min (Cockcroft-Gault) based on Cystatin C
* Tracheostomy or non-invasive ventilation (NIV) use > 22 hours per day
* Inability to swallow tablets
* Contraindication therapy:

  * Allergy for one of the product's active pharmaceutical ingredients (APIs) or excipients.
  * Antihypertensive treatment [Trimetazidine may cause hypotension]
* Evidence of malignant disease
* Significant neuromuscular disease other than ALS/MND
* Ongoing disease that may cause neuropathy
* Pregnancy or breastfeeding
* Females actively seeking to become pregnant who are not using an adequate form of contraceptive as detailed in the Inclusion criteria.
* Deprivation of freedom by administrative or court order

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events; Safety and Tolerability | 16 weeks
  The occurrence of adverse events, as assessed by Common Terminology Criteria for AEs Version 5, during the 12-week on-treatment period and 4-week wash-out period (16 weeks total).
Level of expression of oxidative stress markers in the plasma and/or serum of trial participants | 16 weeks
  Expression of oxidative stress markers (malondialdehyde, 8-hydroxy-2'-deoxyguanosine, interleukin-6; assessed by liquid chromatography-mass spectrometry/mass-spectrometry or multiplexing) in the plasma and/or serum of trial participants throughout the treatment period (12-week) and at the end of the wash-out period (4 weeks)

SECONDARY OUTCOMES:
Level of expression of oxidative stress markers in the plasma and/or serum of trial participants to inform future clinical trials in ALS/MND | 16 weeks
  Assessment of the expression of oxidative stress markers (malondialdehyde, 8-hydroxy-2'-deoxyguanosine, interleukin-6; assessed by liquid chromatography-mass spectrometry/mass-spectrometry or multiplexing) in the plasma and/or serum of trial participants throughout the treatment period (12-week) and at the end of the wash-out period (4 weeks) to determine suitability for incorporation into future trial design

CONTACTS AND LOCATIONS:
Overall Officials: Shyuan Ngo, PhD, Principal Investigator — The University of Queensland; Robert Henderson, MBBS, PhD, Principal Investigator — Royal Brisbane & Women's Hospital; Leonard van den Berg, MD, PhD, Principal Investigator — UMC Utrecht; Ammar Al-Chalabi, MB ChB, PhD, Principal Investigator — King's College London; Frederik Steyn, PhD, Principal Investigator — The University of Queensland; Ruben van Eijk, MD, PhD, Principal Investigator — UMC Utrecht
Locations (3):
- Royal Brisbane & Women's Hospital, Brisbane, Queensland, Australia
- University Medical Centre Utrecht, Utrecht, Netherlands
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No